CLINICAL TRIAL: NCT02104167
Title: An Open-Label Clinical Study of the Safety and Efficacy of the ROI-C Anterior Cervical Interbody Fusion Device Using the VerteBRIDGE Plating System
Brief Title: Retrospective/Prospective Data Collection on the LDR ROIC Interbody Fusion Device With VerteBRIDGE Plating
Status: Completed | Type: Observational
Sponsor: LDR Spine USA (Industry)
Responsible Party: Sponsor
Other Study IDs: ROIC100
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-01

CONDITIONS: Degenerative Disc Disease
Keywords: DDD; degenerative disc disease; cervical spine; fusion rate
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Operated Subjects: ROIC interbody cage with VerteBRIDGE plating
  Interventions: Device: ROIC interbody cage with VerteBRIDGE plating

INTERVENTIONS:
Device: ROIC interbody cage with VerteBRIDGE plating

SUMMARY:
The purpose of this combined retrospective and prospective clinical study is to examine the clinical outcomes of the ROI-C® anterior cervical interbody fusion device with VerteBRIDGE® plating to treat single level degenerative disc disease between C2 and T1 in the short term, with a focus on fusion rates.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have degenerative disc disease (DDD) of the cervical spine with accompanying radicular symptoms at one level between C2 and T1.
* The subject can have the ROI-C device at only one level.
* Autograft must have been used with the ROI-C device.
* Subject should have had a minimum of 6 (six) weeks of non-operative treatment prior to surgery.
* Subject must be at least 21 years of age at the time of surgery

Exclusion Criteria:

* No BMP was used in the interbody cage
* Subject was a prisoner at the time of surgery
* Subject was pregnant at the time of surgery
* Subject had an active infection or sepsis at the time of surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be drawn from community surgeon practices in which the subjects have already received the device and who meet the Inclusion/Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Jackson, MD, Principal Investigator — Orange County Neurosurgical Associates
Locations (7):
- United States (7):
  - Orange County Neurological Associates, Laguna Hills, California
  - Orthpedic Specialists of Northwest Indiana, Munster, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - New England Orthopedic Surgeons, Springfield, Massachusetts
  - St Francis Hospital, Greenville, South Carolina
  - Franciscan Neurosurgery Associates, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Operated Subjects With ROI-C Device: Subjects who were operated on or after Jan. 1, 2011 and who have a minimum of 12 months post-operative time prior to the final study visit.
Period: Overall Study
Arm/Group | Operated Subjects With ROI-C Device
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects who were operated on or after Jan. 1, 2011 and who have a minimum of 12 months post-operative time prior to the final study visit.
Arm/Group | Operated Subjects With ROI-C Device
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fusion
Description: Rate of fusion using A/P, lateral, and flexion/extension radiographs at each time point; defined by the presence of bridging bone with less than 2° segmental motion in flexion/extension and less than 3mm of A/P translation.
Time Frame: 12 months or more after device implantation; mean follow up 20.7 months
Measure: Number; unit: Percentage of Participants
Arm/Group | Operated Subjects With ROI-C Device
Number analyzed (Participants) | 110
Percentage of Participants | 99.1

2. Secondary Outcome: Mean Neck Disability Index (NDI), Visual Analog Scale (VAS)- Neck Pain, Visual Analog Scale (VAS)-Right and Left Arm Pain
Description: NDI is a standard instrument for measuring self-rated disability due to neck pain. It is scored from 0-50, with results multiplied by 2 to arrive at a percentage. Lowest scores represent no disability, high scores represent worse disability. A VAS is a measurement instrument for pain that measures the degree across a continuum or straight line. The endpoints define extreme limits, from 0-10, with 0 representing no pain and 10 severe pain.
Time Frame: 12 months (Last available visit) post surgery
Population: Operated Subjects
Measure: Mean (Full Range); unit: Units on a Scale
Arm/Group | Operated Subjects With ROI-C Device
Number analyzed (Participants) | 110
Units on a Scale
  NDI | 19.0 [0 to 72]
  VAS Neck | 26.5 [0 to 100]
  VAS Left Arm | 15.3 [0 to 89]
  VAS Right Arm | 12.5 [0 to 100]

ADVERSE EVENTS:
Time Frame: Date of surgery through last follow up visit, mean of 20.7 months
Description: Any change from baseline in a subject's condition during the clinical study. This includes events that are related to the device as well as events that are not related to the device.
Arm/Group | Operated Subjects With ROI-C Device
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 2/110
Other Adverse Events (participants affected / at risk) | 42/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operated Subjects With ROI-C Device (N=110)
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operated Subjects With ROI-C Device (N=110)
Upper extremity pain/numbness (Musculoskeletal and connective tissue disorders) | 11 (16)
Fall/Injury (Musculoskeletal and connective tissue disorders) | 10 (12)
Lower back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck Pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Shoulder injury (Musculoskeletal and connective tissue disorders) | 8 (9)

LIMITATIONS AND CAVEATS:
This was a single-arm study that enrolled participants retrospectively. An active control is not available for comparison of results and changes from baseline are not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No